CLINICAL TRIAL: NCT05976997
Title: Prospective, Single Arm, Single Center Study of Duvelisib Combined With Chidamide in the Treatment of Newly Diagnosed Peripheral T-cell Lymphoma (PTCL)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Liling Zhang (Other)
Collaborators: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Liling Zhang, chief physician, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-KBT-PTCL-C01
Record Dates: First submitted 2023-07-16; First posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-07

CONDITIONS: Newly Diagnosed Peripheral T-cell Lymphoma
Keywords: Duvelisib; Chidamide; Peripheral T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — duvelisib; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Duvelisib-Chidamide (Experimental): Patients with newly diagnosed PTCL were treated with a combination of Duvelisib and Chidamide. The dose of Duvelisib was 25mg twice a day. Every 4 weeks (28 days) is a cycle with a total of 2 cycles.
  Interventions: Drug: Duvelisib, Chidamide

INTERVENTIONS:
Drug: Duvelisib, Chidamide — Duvelisib, 25mg, BID, PO; Chidamide, 20mg, BIW, PO;

SUMMARY:
This is a prospective, single arm, single center study to evaluate the efficacy and safety of Duvelisib combined with Chidamide in the treatment of newly diagnosed peripheral T-cell lymphoma.

DETAILED DESCRIPTION:
This is a prospective, single arm, single center study, including two phases. It plans to recruit36 patients with clinically diagnosed primary PTCL who will be treated with Duvelisib and Chidamide. In the first phase Duvelisib is Oral administration at a dose of 25mg twice a day, and every 4 weeks (28 days) was a cycle. Next administration will be depend on whether the efficacy reaches CR in the second phase.

ELIGIBILITY:
Inclusion Criteria:

-

1.Age: 18-70 Years (Contains boundary values 18 and 70);

* 2.The newly diagnosed PTCL confirmed by histopathology is one of the following subtypes;

  a) Angioimmunoblastic T-cell lymphoma (AITL); b) Follicular T helper cell lymphoma (T-FHCL); Including but not limited to the above two subtypes;
* 3.ECOG ≤ 3;
* 4.At least one measurable or evaluable tumor lesion according to the Lugano-2014 standard;
* 5.Expected survival ≥ 3 months;
* 6.Subjects fully understand and voluntarily participate in this study and sign informed consent;

Exclusion Criteria:

-

1.Subjects who have previously received systemic treatment for lymphoma or currently undergoing anticancer treatment;

* 2.Subjects with central nervous system (CNS) lymphoma or lymphoma involving CNS;
* 3.Significant active heart disease within the past 6 months, including: New York Heart Association (NYHA) Class III/IV congestive heart failure unstable angina pectoris or angina requiring surgical or medication intervention, and/or myocardial infarction;
* 4.Uncontrolled systemic fungal, bacterial, or viral infections (defined as persistent signs/symptoms related to infection that have not improved despite the use of appropriate antibiotics, antiviral therapy, and/or other treatments);
* 5.Human immunodeficiency virus (HIV), hepatitis B or hepatitis C infection and history of severe skin reaction;
* 6.Subjects with any other active malignant tumor at the time of screening, except for adequately treated cervical Carcinoma in situ or breast cancer Carcinoma in situ, skin Basal-cell carcinoma or local skin squamous cell carcinoma;
* 7.Pregnant women, lactating women, patients who refused to take effective contraceptive measures during the study;
* 8.Any serious uncontrolled systemic disease;
* 9.increasing the risk of the subject or interfering with the test results determined by the investigator;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Safety: Hematologic and non-hematologic toxicities (NCI CTCAE v5.0) | from the initiation of the first dose to 28 days after the last dose
  To identify the incidence of AE and SAE in clinical trial

SECONDARY OUTCOMES:
Objective response rate (ORR) | up to 26 weeks
  To evaluate the efficacy of anti-lymphoma
Complete remission rate (CR) | up to 26 weeks
  To evaluate the efficacy of anti-lymphoma
Duration of Response（DOR） | The time from the first assessment as CR or PR to the first assessment as PD or death (due to any cause)，assessed up to 12 months
  To evaluate the efficacy of anti-lymphoma
Progression free survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 20 months
  To evaluate the efficacy of anti-lymphoma
Overall survival (OS) | From date of randomization until the date of death from any cause, assessed up to 20 months
  To evaluate the efficacy of anti-lymphoma

CONTACTS AND LOCATIONS:
Overall Officials: Liling Zhang, M.D, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China